CLINICAL TRIAL: NCT01237652
Title: Perioperative Myocardial Ischemia in Isolated Systolic Hypertension (PROMISE)
Brief Title: Perioperative Myocardial Ischemia in Isolated Systolic Hypertension
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Ashraf Fayad, The Ottawa Hospita, University of Ottawa
Other Study IDs: ESA 5971
Record Dates: First submitted 2010-10-13; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension; Myocardial Ischemia
Keywords: Isolated Systolic Hypertension; Perioperative Myocardial Ischemia; Perioperative Cardiovascular adverse events
MeSH Terms: conditions — Hypertension; Myocardial Ischemia; Isolated Systolic Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ISH and normotensive: This is a prospective cohort study to compare the incidence of perioperative myocardial ischemia between ISH and normotensive patients admitted for elective non-cardiac surgery. To reduce the number of confounding factors for perioperative myocardial ischemia, RCRI Class I or II patients will be recruited.
- ISH, Normotensive: This is a prospective cohort study to compare the incidence of perioperative myocardial ischemia between ISH and normotensive patients admitted for elective non-cardiac surgery. To reduce the number of confounding factors for perioperative myocardial ischemia, RCRI Class I or II patients will be recruited.

SUMMARY:
During or after surgery, patients may suffer heart attacks or other heart complications, increasing the hospital stay by 11 days on average and costing an estimated US$20 billion in 1990.Many risk factors have been identified but there are no properly conducted studies to look at Blood pressure (BP) as a risk factor around the time of surgery. The investigators believe there is a good possibility that systolic BP (SBP) is a risk factor but currently unrecognized. When measuring BP, two numbers are obtained. The upper number is called SBP and a lower number called diastolic BP (DBP). If the numbers are high, this means that the patient has a high BP or hypertension. If the SBP is high while DBP is normal, it is called isolated systolic hypertension (ISH)> ISH is increasingly recognized as a major risk factor for heart problems. The relationship between ISH and heart complications around the time of surgery is poorly understood. Previous studies did not look at such a relationship. Because of that, there are no guidelines for ISH management at the time of surgery. Generally, these patients go through surgery as if they have no increased risk. Studies are starting to show that the bulk of these heart complications happen in patients thought to have low risk factors not yet identified, including ISH.

The investigators believe that the oxygen supply to the heart can be compromised around the time of surgery in ISH patients Chemicals known as stress hormones are secreted around the time of surgery, increasing oxygen needs in the heart and may make the oxygen supply to the heart muscle critical (know as myocardial ischemia). This in turn may result in a heart attack and death. Studies have shown that patients with myocardial ischemia stand a 9-fold increase in odds ratio of suffering a heart attack, worsening of angina, or death.

This study aims to compare the incidence of myocardial ischemia in patients with ISH and normal BP patients around the time of surgery using a special heart monitor. In addition, the study aims to determine the prevalence of ISH among surgical patients and to document complications like heart attacks, heart failure, stroke and death after surgery.

This research project will be conducted at the Ottawa Hospital by a multi-disciplinary research group (perioperative research group)which includes anesthesiology, cardiology, general surgery and epidemiology. The research group secured HSFO funding for this study.

DETAILED DESCRIPTION:
Ethics approval is already obtained. Consented patients will be screened for ISH in the pre-surgical clinic, utilizing BP automated machine. Patients with ISH or normal diastolic function (control group) will be enrolled. During and after surgery, they will be monitored for changes consistent with myocardial ischemia. A special heart monitor, called ambulatory ECG monitor (Holter monitor), will be used to record, document and count any episodes of myocardial ischemia. A designated research coordinator will be assigned to the study for the recruitment, screening, daily tracking and data collection. The heart monitoring for each patient in the study will be reviewed by the research group. Data will be collected and analysed.

This is the first study looking exclusively at ISH as a risk factor around the time of surgery. Studies suggest that investigators may be labelling surgical patients at risk of a heart attack as "low risk" when in fact the bulk of those heart attacks are in patients labeled "low risk". The finding that ISH patients have a higher incidence of myocardial ischemia will provide evidence for the next level of research. If ISH is in fact a risk factor for heart attacks around the time of surgery, the investigators will identify a group of patients in whom the investigators can lower this risk by instituting appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* ISH or normotensive (as per Patient Recruitment and Informed Consent section)
* Elective non cardiac surgical procedure
* Expected to stay in hospital ≥ 48 hours
* Revised cardiac risk index (RCRI) ≤ 251

Exclusion Criteria:

* Atrial fibrillation
* Left bundle branch block (LBBB)
* Myocardial infarction < 3 months
* Decompensated congestive heart failure
* Unstable coronary syndrome
* Dialysis
* Emergency surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perioperative ISH and normotensive presenting for Non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Incidence of perioperative myocardial ischemia in ISH patients | 48 hours postop
  To determine if the incidence of perioperative myocardial ischemia in ISH patients is triple that of normotensive patients admitted for non-cardiac surgery, as determined by 48-hour ambulatory ST segment ECG monitoring.

SECONDARY OUTCOMES:
Proportion of ISH Patients admitted for non-cardiac surgery | day of surgery
  To determine the proportion of patients admitted for non-cardiac surgery with treated and untreated Isolated Systolic Hypertension, normotension, and systemic hypertension with diastolic elevation;
Determine the demographics of patients admitted for non-cardiac surgery with Isolated Systolic Hypertension | day of surgery
  Demographics include age, diabetes, ASA status.
To determine the overall incidence of perioperative MI, Cardiovascular death, cardiac arrests, or CVA in RCRI Class I or II patients admitted for non cardiac surgery | 1 week
  Outcomes and complications data are collected from the day of surgery until discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Fayad, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Fayad AA, Yang HY, Ruddy TD, Watters JM, Wells GA. Perioperative myocardial ischemia and isolated systolic hypertension in non-cardiac surgery. Can J Anaesth. 2011 May;58(5):428-35. doi: 10.1007/s12630-011-9477-7. Epub 2011 Feb 24. PMID 21347737